CLINICAL TRIAL: NCT06282549
Title: A Prospective Long-term Cohort Study to Identify the Predictive Model of Cardiocerebrovascular Risk Factors in Elderly Patients with More Than Three Antihypertensive Agents in Patients with Essential Hypertension in Korea
Brief Title: Study to Evaluate the Efficacy and Safety of TEL/AML/CTD in Elderly Patients with Essential Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YMC046
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Essential Hypertension
Keywords: Telmisartan/Amlodipine/Chlorthalidone Fixed-Dose Combination (Truset)
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Telmisartan/Amlodipine/Chlorthalidone(Truset) — Telmisartan/Amlodipine/Chlorthalidone 40/5/12.5 mg or Telmisartan/Amlodipine/Chlorthalidone 80/5/12.5 mg or Telmisartan/Amlodipine/Chlorthalidone 80/5/25 mg

SUMMARY:
This study is to develop a predictive model for cardiocerebrovascular risk factors in elderly patients with essential hypertension with Telmisartan, Amlodipine, and Chlorthalidone Fixed-Dose Combination.

DETAILED DESCRIPTION:
This is a phase IV, open-label, prospective, long-term cohort, observational study to identify the predictive model of cardiocerebrovascular risk factors in elderly patients with more than three antihypertensive agents in patients with essential hypertension in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. A patient over 65-year-old with essential hypertension
2. A patient with essential hypertension who require treatment with 3 or more antihypertensive medication, as determined by investigator's decision
3. A patient with no MACCE within 6 months prior to the enrollment
4. A patient who voluntarily signed the informed consent form

Exclusion Criteria:

1. A patient who participates in clinical trial
2. A patient who are contraindicated for the Truset tablet according to the label.
3. A patient who is unable to complete the study judged by the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients in General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1219 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of MACCE(Major Adverse Cardiovascular and Cerebrovascular Events) | 12, 24 and 36months
  Percentage of MACCE(Major Adverse Cardiovascular and Cerebrovascular Events) after treatment at 12, 24 and 36months if applicable

SECONDARY OUTCOMES:
Percentage of MACCE(Major Adverse Cardiovascular and Cerebrovascular Events) in patients with asymptomatic target organ damage | 12, 24 and 36months
  Percentage of MACCE(Major Adverse Cardiovascular and Cerebrovascular Events) in patients with asymptomatic target organ damage after treatment at 12, 24 and 36months if applicable
Mean Systolic Blood Pressure (MSBP)/ Diastolic Blood Pressure (MDBP) | 12, 24 and 36months
  To evaluate change from baseline in Mean Systolic Blood Pressure (MSBP)/ Diastolic Blood Pressure (MDBP) measured by the Institution at 12, 24 and 36months if applicable
Patients Achieving the treatment goal in Mean Systolic Blood Pressure (MSBP) | 36months
  To evaluate the percentage of patients who reached the treatment goal for Mean Sitting Blood Pressure (MSBP) < 140/90 mmHg measured by the Institution at 12, 24 and 36months if applicable
Percentage of patients who terminated the treatment | 36months
  To evaluate the percentage of patients who terminated the treatment before 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Lee, Principal Investigator — Veterans Health Service Medical Center
Locations (5):
- South Korea (5):
  - Busan Veterans Hospital, Busan
  - Daegu Veterans Hospital, Daegu
  - Gwangju Veterans Hospital, Gwangju
  - Konkuk University Medical Center, Seoul
  - Veterans Health Service Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No